CLINICAL TRIAL: NCT06967870
Title: The Effect of Cranial Osteopathy Intervention on Sensory Profile, Sleep Quality, Colic Symptoms and Motor Movements in Preterm Babies
Brief Title: The Effect of Cranial Osteopathy Intervention in Preterm Babies
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Eylem TÜTÜN YÜMİN, Professor, Abant Izzet Baysal University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AIBU-FTR-ETY-04
Record Dates: First submitted 2025-03-03; First posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Osteopathy; PreTerm Neonate; Sensory Profiles; Colic; Sleep Quality; Motor Development of Premature Infants
Keywords: manual therapy; premature; sensory integration; early intervention; cranial
MeSH Terms: conditions — Colic; Sleep Initiation and Maintenance Disorders; Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Osteopathy intervention group (Experimental): Beginning of the project assesment will be made, home exercises are going to be explained and said to continue exercises every day. Cases in this group will take 6 osteopathy sessions weekly. After 6 weeks assesment will be made again.
  Interventions: Other: Osteopathic intervention; Other: Home based exercise education
- Home based exercises group (Active Comparator): Beginning of the project assesment will be made, home exercises are going to be explained and said to continue exercises every day. After 6 weeks assesment will be made again.
  Interventions: Other: Home based exercise education

INTERVENTIONS:
Other: Osteopathic intervention — Researcher will use osteopathic techniques on cranial area includes light touch.
  Home based exercises will be show on cases and demand to do exercise regularly
  Arms: Osteopathy intervention group
Other: Home based exercise education — Home based exercises will be show on cases and demand to do exercise regularly.

SUMMARY:
There are planing to have 2 groups of premature born cases. Each group will include 15 cases. Participants are need to be 28-37 weeks born and no older than post term 6 weeks. All cases are going to be evaluated. Home based exercise plan is going to be explained. The experimental group is going to take 6 osteopathic sessions weekly. After 6 weeks cases are going to be evaluated again.

DETAILED DESCRIPTION:
Babies born at or before the 37th week of pregnancy are defined as preterm babies. While the number of premature babies has increased in recent years, the survival rates of preterm babies have also increased with the development of neonatal intensive care units. Neurodevelopmental problems can be seen at a higher rate in premature babies compared to term babies. In preterm births, birth occurs at critical stages of brain and nervous system development in the baby. It has been stated in the literature that even late preterm babies may experience problems in sensory processing and regulation stages. The addition of factors such as neonatal intensive care history to preterm birth causes them to score even lower in terms of sensory profile compared to term babies. It has been stated that preterm babies are in the high-risk group in terms of sensory processing problems. In a systematic review conducted in 2019, it was stated that premature babies and children have sensory modulation problems at a rate of 28-87%; sensory processing problems at a rate of 9-70%, and sensory-based motor processing problems at a rate of 20-70%.

Colic in babies; It is a condition characterized by sudden, persistent and restless crying in a generally healthy situation. Abdominal bloating and irritability often accompany the crying. It is difficult for the baby to calm down and fall asleep.Although the etiopathogenesis of colic in the neonatal period has not been fully determined, it has been stated that the underdeveloped nervous system, gastrointestinal system and stress factors are triggers. Studies have shown that the frequency of colic increases as the baby's gestational age decreases.

Sleep is the primary activity of the developing brain in early life, so it is not surprising that sleep plays a very important role in brain development. The existence of a sleep-wake cycle, sleep architecture and the percentage of the 24-hour period spent sleeping in the neonatal period have been associated with neurodevelopmental outcomes.

The importance of early intervention in preterm babies is emphasized in the literature. Although there are no protocol-determined intervention methods for babies in the developmental risk group, it has been recommended to start developmental intervention as early as possible. Osteopathic manual therapy applications consist of drug-free, non-invasive, and manually applied methods. They are important methods used to contribute to the health of babies. The focus is on tissue tensions that occur especially in the cranial regions of babies. There are a limited number of studies in the literature on the effectiveness of cranial osteopathic applications. No study has been found on the effect of cranial osteopathy on the sensory profile of the baby. Although there are studies evaluating the relationship between the baby's sleep quality and colic symptoms, different results have been obtained. This study was planned to contribute to the literature by investigating the effect of cranial osteopathy on the sensory profile, sleep quality and colic symptoms in premature babies. In the study, in addition to obtaining evidence-based data on cranial osteopathic applications, it was aimed to examine the effects on the sensory profile, sleep quality, colic symptoms and motor performance of preterm babies.

ELIGIBILITY:
Inclusion Criteria:

* Premature birth (<37 weeks)
* Corrected age <6 weeks.
* Discharged to home
* Stable condition
* Family agrees to continue home program

Exclusion Criteria:

* Having a congenital cyanotic heart problem,
* Being born earlier than 28 weeks,
* The family not accepting to participate in the study,
* Neglecting check-ups and sessions,
* Using a respiratory appliance,
* Presence of craniosynostosis,
* Being included in another physiotherapy program during the study period

Ages: 1 Week to 6 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2025-05-05 (Estimated); Primary Completion 2025-08-28 (Estimated); Study Completion 2025-10-08 (Estimated)

PRIMARY OUTCOMES:
Test of Infant Motor Performance | 6 weeks
  The test is a motor outcome measure designed to assess posture and selective control of movement in infants for functional performance in daily life. The test consists of 31 items in standard format, 28 of which are made by observing spontaneous activities and scoring them as pass or fail. Getting higher points means better motor control.

SECONDARY OUTCOMES:
Assessment of General Movements | 6 weeks
  This is a diagnostic tool for the functional assessment of the young nervous system. General Movements is a diagnostic tool based on visual gestalt perception of videoed agespecific normal or abnormal general movements. Motor Optimality Scores < = 23 at 14-16 weeks of corrected age are predictive of motor, cognitive, and neurosensory motor impairment, and scores <=15 are predictive of CP.
The Infant Colic Scale | 6 weeks
  This Scale was developed to help diagnose colic. The scale has a total of 22 items in 5 subscales. Cow's milk/soy protein allergy/intolerance, immature gastrointestinal system, immature central nervous system, difficult baby temperament, parent-baby interaction-problem baby. Infant colic scale items are evaluated over 6 points. Likert-type scale is used. Low score is an indicator of colic
Brief Infant Sleep Questionnaire | 6 weeks
  It is a questionnaire that provides objective measurement of infant sleep. It has 13 items. It is an assessment form regarding sleep patterns, sleep ecology and parents' sleep perceptions of babies aged 0-36 months. The questionnaire includes specific items about the baby's day and night sleep patterns as well as sleep-related behaviors and parental perception.

CONTACTS AND LOCATIONS:
Locations (1):
- Bahriye Baş, Bursa, Osmangazi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No